CLINICAL TRIAL: NCT01256385
Title: A T1 Translational Multicenter Randomized Phase II Study of Temsirolimus Versus Cetuximab Plus Temsirolimus in Patients With Recurrent / Metastatic Head and Neck Cancer, Who Failed Prior EGFR Based Therapy
Brief Title: Temsirolimus With or Without Cetuximab in Patients With Recurrent and/or Metastatic Head and Neck Cancer Who Did Not Respond to Previous Therapy
Acronym: MAESTRO HN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02596; NCI-2011-02596 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000689896; UCCRC-10-428-B; 10-428-B; 10-428-B (Other: University of Chicago Comprehensive Cancer Center P2C); 8692 (Other: CTEP); N01CM00071 (NIH); N01CM00099 (NIH); N01CM62201 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Laryngeal Verrucous Carcinoma; Recurrent Lip and Oral Cavity Squamous Cell Carcinoma; Recurrent Metastatic Squamous Cell Carcinoma in the Neck With Occult Primary; Recurrent Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Recurrent Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Recurrent Oral Cavity Verrucous Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Recurrent Salivary Gland Carcinoma; Salivary Gland Squamous Cell Carcinoma; Squamous Cell Carcinoma Metastatic in the Neck With Occult Primary; Stage IV Hypopharyngeal Squamous Cell Carcinoma; Stage IV Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage IVA Laryngeal Squamous Cell Carcinoma; Stage IVA Laryngeal Verrucous Carcinoma; Stage IVA Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVA Major Salivary Gland Carcinoma; Stage IVA Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVA Oral Cavity Verrucous Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Stage IVB Laryngeal Squamous Cell Carcinoma; Stage IVB Laryngeal Verrucous Carcinoma; Stage IVB Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVB Major Salivary Gland Carcinoma; Stage IVB Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVB Oral Cavity Verrucous Carcinoma; Stage IVB Oropharyngeal Squamous Cell Carcinoma; Stage IVC Laryngeal Squamous Cell Carcinoma; Stage IVC Laryngeal Verrucous Carcinoma; Stage IVC Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVC Major Salivary Gland Carcinoma; Stage IVC Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVC Oral Cavity Verrucous Carcinoma; Stage IVC Oropharyngeal Squamous Cell Carcinoma; Tongue Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphoid Interstitial Pneumonia; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — Cetuximab; temsirolimus; Sirolimus

ARMS (2):
- Arm A (cetuximab and temsirolimus) (Experimental): Patients receive temsirolimus IV over 30-60 minutes and cetuximab IV over 1-2 hours once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Other: Laboratory Biomarker Analysis; Drug: Temsirolimus
- Arm B (temsirolimus) (Experimental): Patients receive temsirolimus as in Arm A. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may cross over to Arm A.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Temsirolimus

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm A (cetuximab and temsirolimus)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase II trial studies how well giving temsirolimus together with cetuximab works compared to temsirolimus alone in treating patients with recurrent and/or metastatic head and neck cancer who did not respond to previous therapy. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving temsirolimus together with cetuximab is more effective than giving temsirolimus alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Primary endpoint is progression free survival (PFS) of cetuximab/temsirolimus combination cohort (Arm A) compared to temsirolimus alone (Arm B).

SECONDARY OBJECTIVES:

I. Progression-free survival (PFS) of cetuximab/temsirolimus combination group (Arm A) and temsirolimus control group (Arm B) compared to a historic control cohort.

II. Subgroup analysis of myofibroblast (+) cohort (PFS). III. Overall survival (OS). IV. Toxicities. V. Response (Response Evaluation Criteria in Solid Tumors [RECIST])/absolute tumor shrinkage (waterfall plot analysis).

VI. Activity of combination therapy (temsirolimus/cetuximab) after failure (progressive disease [PD]) of temsirolimus monotherapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive temsirolimus intravenously (IV) over 30-60 minutes and cetuximab IV over 1-2 hours once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive temsirolimus as in Arm A. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may cross over to Arm A.

After completion of study therapy, patients are followed up for a minimum of 8 weeks and then once a year for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed diagnosis of squamous cell carcinoma of head and neck origin not amenable to curative intent therapy; information on prior exposure to cetuximab (duration, single agent/combined with chemotherapy/combined with radiation, best response, interval prior to study entry) will be collected
* Progressive disease by RECIST criteria (or unequivocal clinical progression) on a cetuximab based therapy in any line of therapy for recurrent/metastatic disease; prior use of cetuximab for recurrent/metastatic disease is defined as palliative intent use either alone or in combination with chemotherapy with a minimum of 2 weeks of uninterrupted treatment with cetuximab; treatment with cetuximab during radiotherapy or chemoradiotherapy is not sufficient
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1
* Presence of measurable lesions by RECIST: patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Knowledge of the anatomic site of the original tumor (oropharynx versus non-oropharynx) or alternatively human papilloma virus (HPV) status; the trial will stratify patients by oropharynx versus non-oropharynx origin; HPV(+) tumors will be counted in the oropharynx cohort, HPV(-) tumors in the non-oropharynx cohort; at a later point all patients will undergo HPV testing as part of this trial; any widely used form of HPV testing is acceptable (including but not limited to HPV in situ hybridization [ISH], p16 testing [immunohistochemistry (IHC)], HPV16 testing, polymerase chain reaction [PCR], hybrid capture, etc)
* Availability of formalin-fixed, paraffin-embedded (FFPE) tissue and blood

  * FFPE: >=14 slides containing tumor, 18 recommended

    * 7-10 slides 5 um thick, AND 7-10 slides 10 um thick, and cut with a clean blade (use new blade if possible or clean vigorously to avoid RNA/DNA, RNase contamination)
  * Blood: two 10 cc ethylenediaminetetraacetic acid (EDTA) purple top tubes (blood); two 2 ml cryovials (serum)
* Patients with human immunodeficiency virus (HIV), not requiring highly active antiretroviral treatment (HAART) therapy are eligible
* Life expectancy of greater than 8 weeks
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits (unless proven Gilbert's disease, which after principal investigator [PI] approval patient may be included)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within 1.5 X normal institutional limits
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document
* Fasting glucose of =< 120 mg/dl and glycosylated hemoglobin (HbA1c) =< 7.5%

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known, active brain metastases should be excluded from this clinical trial; patients with treated brain metastases stable for >= 12 weeks are eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temsirolimus or cetuximab
* Concurrent life-threatening diseases: patients with diseases which with reasonable certainty do not limit life expectancy to 12 months or less are eligible; assessment of such concurrent illnesses should be by the principal investigator
* Use of strong inhibitors/inducers of CYP3A4 is not permitted
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study
* Breastfeeding should be discontinued if the mother is treated with temsirolimus
* HIV-positive patients with normal immune function (CD4 count > 200) are eligible if there are no drug interactions with temsirolimus or cetuximab; patients with impaired immune function are ineligible due to the risk of additional immunosuppression from temsirolimus therapy
* Concurrent administration of temsirolimus with vaccinations is to be avoided and a 14-day window from administration of the vaccine is advised; in emergent situations this policy may be revisited by the PI if deemed important for the patient's health
* Poorly controlled hyperglycemia (HbA1C > 7.5%) or hyperlipidemia are exclusion criteria; hyperglycemia or hyperlipidemia need to be appropriately managed and controlled
* Concurrent use of warfarin is allowed, but requires close monitoring of prothrombin time (PT)/international normalized ratio (INR)
* Patients with clinically significant pneumonitis/pulmonary infiltrates unless there is a known and treatable cause for the condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, Principal Investigator — University of Chicago Comprehensive Cancer Center P2C
Locations (24):
- United States (23):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus)
Started | 43 | 43
Crossover From Arm B to Arm A | 0 | 15
Completed | 40 | 40
Not Completed | 3 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: Three patients from each treatment arm did not start treatment and are considered non-evaluable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Full Range); unit: years] | 63 [48 to 86] | 63 [39 to 81] | 63 [39 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 32 | 37 | 69
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression determined using RECIST criteria: >=20% increase in the sum of the longest diameters of target lesions from nadir, occurrence of new lesions, or progression of non-target lesions.
Time Frame: From start of treatment to time of progression or death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus)
Number analyzed (Participants) | 40 | 40
days | 105 [70 to 136] | 105 [77 to 147]
Statistical Analysis 1: Comparison: Arm A (Cetuximab and Temsirolimus) vs Arm B (Temsirolimus); Test type: Superiority or Other; p = 0.73, Log Rank

2. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization until death from any cause
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus)
Number analyzed (Participants) | 40 | 40
days | 177 [146 to 247] | 176 [131 to 316]
Statistical Analysis 1: Comparison: Arm A (Cetuximab and Temsirolimus) vs Arm B (Temsirolimus); Test type: Superiority or Other; p = 0.87, Log Rank

3. Secondary Outcome: Overall Response Rates (OR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Statistics reported are for Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus)
Number analyzed (Participants) | 40 | 40
percentage of participants | 12.5 [4.2 to 26.8] | 2.5 [0.1 to 13.2]
Statistical Analysis 1: Comparison: Arm A (Cetuximab and Temsirolimus) vs Arm B (Temsirolimus); Test type: Superiority or Other; p = 0.20, Fisher Exact

4. Secondary Outcome: PFS vs. Historical Control Cohort
Description: PFS at 4 months in Arm A and Arm B will each be compared with a 4-month historical control rate of 21.4%. The historical data appears in two publications, an ASCO abstract: Abidoye, ASCO Annual Meeting 2006: 5568 and de Souza, Davis, et al, Clin Cancer Res 2012; 18(8):2336-2343.
Time Frame: From start of treatment to time of progression or death of any cause, assessed at 4 months
Population: Note: Each arm is separately compared to an historical rate of 21.4%, based on a one-sided test at the 0.05 significant level. Since the 90% CIs each exclude 21.4%, the 4-month PFS rate in both arms exceeds the fixed historical control rate.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus)
Number analyzed (Participants) | 40 | 40
percentage of participants | 41.3 [28.3 to 54.3] | 36.4 [22.6 to 50.2]
Statistical Analysis 1: Comparison: Arm A (Cetuximab and Temsirolimus); PFS at 4 months in Arm A was compared with a 4-month historical control rate of 21.4%, using a one-sided test at the 0.05 significant level. The historical data appear in two publications, an ASCO abstract: Abidoye, ASCO Annual Meeting 2006: 5568, and de Souza, Davis, et al, Clin Cancer Res 2012; 18(8):2336-2343 (see Figure 1); Test type: Superiority; p = 0.006, Chi-squared
Statistical Analysis 2: Comparison: Arm B (Temsirolimus); PFS at 4 months in Arm B was compared with a 4-month historical control rate of 21.4%, using a one-sided test at the 0.05 significant level. The historical data appear in two publications, an ASCO abstract: Abidoye, ASCO Annual Meeting 2006: 5568, and de Souza, Davis, et al, Clin Cancer Res 2012; 18(8):2336-2343 (see Figure 1); Test type: Superiority; p = 0.037, Chi-squared — 1-sided

5. Secondary Outcome: Grade 3 or Higher Hematological Toxicity
Description: Incidence of hematological toxicities at least possibly related to study drug, graded based on Common Terminology Criteria for Adverse Events version 4
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus)
Number analyzed (Participants) | 40 | 40
percentage of participants | 17.5 [7.3 to 32.8] | 25 [12.7 to 41.1]
Statistical Analysis 1: Comparison: Arm A (Cetuximab and Temsirolimus) vs Arm B (Temsirolimus); Test type: Superiority or Other; p = 0.59, Fisher Exact

6. Secondary Outcome: Percentage of Responses After Crossover From Control Arm to the Combination Arm, Assessed According to RECIST
Description: Percentage of responses (if any) after crossover from the control arm to the combination arm will be evaluated qualitatively. This is includes complete and partial responses, and is different from Outcome Measure 8 below, which includes complete and partial responses as well as stable disease.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus)
Number analyzed (Participants) | 0 | 15
percentage of participants |  | 0 [0 to 21.8]

7. Secondary Outcome: PFS of Myofibroblast (+) Cohort
Time Frame: From start of treatment to time of progression or death of any cause, assessed up to 5 years
Population: Myofibroblast status was not determined. Concerns about the validity/technical feasibility as well as availability of the assay led us to decide to not perform the assay. We do not intend to perform this assay anymore.
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Responses/Disease Stabilization for Patients Crossing Over to the Combination Therapy After Progressing on Arm B.
Description: Assessed according to RECIST. This is includes complete and partial responses as well as stable disease, and is different from Outcome Measure 6 above, which includes only complete and partial responses.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus)
Number analyzed (Participants) | 0 | 15
percentage of participants |  | 26.7 [7.8 to 55.1]

ADVERSE EVENTS:
Arm/Group | Arm A (Cetuximab and Temsirolimus) | Arm B (Temsirolimus)
Serious Adverse Events (participants affected / at risk) | 14/40 | 19/40
Other Adverse Events (participants affected / at risk) | 39/40 | 37/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Cetuximab and Temsirolimus) (N=40) | Arm B (Temsirolimus) (N=40)
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2
Anorectal infection (Infections and infestations) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Death NOS (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Edema face (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 1 | 1
General disorders and administration site conditions - Other (General disorders) | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hypernatremia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 3 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural infection (Infections and infestations) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Scrotal infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Wound infection (Infections and infestations) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Cetuximab and Temsirolimus) (N=40) | Arm B (Temsirolimus) (N=40)
Alanine aminotransferase increased (Investigations) | 11 | 10
Alkaline phosphatase increased (Investigations) | 10 | 7
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Anemia (Blood and lymphatic system disorders) | 24 | 26
Anorexia (Metabolism and nutrition disorders) | 11 | 15
Anxiety (Psychiatric disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Aspartate aminotransferase increased (Investigations) | 9 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Blurred vision (Eye disorders) | 2 | 1
CD4 lymphocytes decreased (Investigations) | 3 | 0
Chills (General disorders) | 3 | 2
Cholesterol high (Investigations) | 9 | 10
Constipation (Gastrointestinal disorders) | 14 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Creatinine increased (Investigations) | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Depression (Psychiatric disorders) | 1 | 8
Diarrhea (Gastrointestinal disorders) | 10 | 5
Dizziness (Nervous system disorders) | 5 | 4
Dry mouth (Gastrointestinal disorders) | 4 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 3
Dysgeusia (Nervous system disorders) | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 5 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Ear pain (Ear and labyrinth disorders) | 1 | 2
Edema face (General disorders) | 7 | 6
Edema limbs (General disorders) | 4 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Eye disorders - Other (Eye disorders) | 2 | 1
Facial pain (General disorders) | 2 | 3
Fatigue (General disorders) | 28 | 30
Fever (General disorders) | 7 | 8
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 2
Headache (Nervous system disorders) | 7 | 7
Hearing impaired (Ear and labyrinth disorders) | 0 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 18 | 19
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypertension (Vascular disorders) | 3 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 8 | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 12 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 15 | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 22 | 2
Hyponatremia (Metabolism and nutrition disorders) | 5 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 12 | 8
Hypotension (Vascular disorders) | 2 | 1
INR increased (Investigations) | 0 | 3
Infections and infestations - Other (Infections and infestations) | 5 | 5
Insomnia (Psychiatric disorders) | 7 | 7
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2
Lung infection (Infections and infestations) | 0 | 2
Lymphedema (Vascular disorders) | 1 | 2
Lymphocyte count decreased (Investigations) | 14 | 17
Mucositis oral (Gastrointestinal disorders) | 16 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Nail infection (Infections and infestations) | 3 | 0
Nausea (Gastrointestinal disorders) | 15 | 14
Neck edema (General disorders) | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Neutrophil count decreased (Investigations) | 3 | 4
Non-cardiac chest pain (General disorders) | 1 | 7
Oral dysesthesia (Gastrointestinal disorders) | 2 | 3
Oral pain (Gastrointestinal disorders) | 5 | 1
Pain (General disorders) | 7 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 1
Papulopustular rash (Infections and infestations) | 2 | 2
Paronychia (Infections and infestations) | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 6
Platelet count decreased (Investigations) | 16 | 14
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 19 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 5
Sinusitis (Infections and infestations) | 0 | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 | 1
Skin infection (Infections and infestations) | 6 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Urinary frequency (Renal and urinary disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 7 | 6
Weight loss (Investigations) | 8 | 8
White blood cell decreased (Investigations) | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less